CLINICAL TRIAL: NCT03256006
Title: Per Effort Study of Inflammation During a 100 Miles
Brief Title: Study Inflammation During a 100 Miles
Acronym: TRAIL PHYSIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Romain Jouffroy, Principal Investigator, Hôpital Necker-Enfants Malades
Other Study IDs: 2017-A02397-46
Record Dates: First submitted 2017-08-10; First posted 2017-08-21 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Response
Keywords: sport exercise; ultra endurance
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pro and anti inflammatory biomarkers (reactive oxygen species)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — Blood sample to study per and post effort evolution markers of systemic inflammation

SUMMARY:
To study per and post effort variations of inflammatory biological markers during a 100 miles

ELIGIBILITY:
Inclusion Criteria:

* adults (age>18years)
* completion of an ultra endurance race (50 miles) during the 2 years before

Exclusion Criteria:

* female
* age<18years

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-10-18 (Estimated); Primary Completion 2018-10-18 (Estimated); Study Completion 2018-10-29 (Estimated)

PRIMARY OUTCOMES:
Variation per and post effort of interleukin 1 plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of interleukin 1 will be measured
Variation per and post effort of interleukin 6 plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of interleukin 6 will be measured
Variation of per and post effort of protein C reactive | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of protein C reactive will be measured
Variation per and post effort of interleukin Tumor Necrosis Factor alpha | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of tumor necrosis alpha will be measured
Variation per and post effort of interleukin 4 plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of interleukin 4 will be measured
Variation per and post effort of interleukin 10 plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of interleukin 10 will be measured
Variation per and post effort of interleukin 13 plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of interleukin 13 will be measured
Variation per and post effort of interleukin tumor growth factor beta plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of tumor growth factor beta
Variation per and post effort of lipids plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of lipids
Variation per and post effort of lipoproteins plasma level | Change measures : departure, 25, 49, 72, 100, 126, 144, 164 kilometers (arrival) then at day 1, day 2 and day 7 after the completion of the race
  Plasma level of per and post effort of lipoproteins

IPD SHARING:
Plan to Share IPD: Undecided